CLINICAL TRIAL: NCT04612322
Title: A Multicenter Registry on the Diagnosis of Patients With Chronic Angina and no Angiographic Coronary Artery Stenosis
Brief Title: MICRO: a Registry Study in Patients With Microvascular Angina
Acronym: MICRO
Status: Recruiting | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Tommaso Gori, Clinical Professor, Johannes Gutenberg University Mainz
Other Study IDs: 2020-2
Record Dates: First submitted 2020-10-10; First posted 2020-11-02 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Microvascular Disease
Keywords: Coronary artery disease; Angina
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing coronary microvascular function assessment
  Interventions: Device: Assessment of microvascular function with intracoronary hemodilution

INTERVENTIONS:
Device: Assessment of microvascular function with intracoronary hemodilution — The pressure/temperature wire allows assessing coronary flow reserve, intracoronary pressure, and coronary flow to calculate multiple parameters of coronary macro- and microvascular function.

SUMMARY:
The evidence above demonstrates that microvascular dysfunction is an important determinant of patient prognosis, which however remains poorly classified. Given the high burden of disease and the severity of the functional impairment in these patients, the lack of a clear definition for this disease has a potentially large clinical importance. It is important to better describe the phenotype of these patients, identify the predictors of prognosis, and determine the impact of diagnosis.

DETAILED DESCRIPTION:
The study is designed as prospective registry. Patients with angina CCS II-IV undergoing assessment of microvascular function will be enrolled.

The study does not interfere with the medical standards at the sites with regards to patient treatment or follow-up care.

Study duration and schedule The duration of this study is expected to be 7 years. The subject recruitment is planned to start in January 2020 and end in January 2022. The actual overall study duration or subject recruitment period may differ from these time periods. Per-patient, the duration of participation will be up to 5 years. Patients will be evaluated at hospital discharge, at 12 months and 5 years (the latter two as telephone contacts).

Number of subjects and study centers It is planned to enroll 1000 subjects in the registry based on power calculations as described. Recruitment and treatment of subjects is expected to be performed in 10 study centers.

Primary endpoint The primary endpoint is the composite of cardiovascular death, myocardial infarction, rehospitalization for angina or heart failure, and unplanned coronary angiography at 12 months.

Secondary endpoints Each of the components of the primary endpoint Seattle Angina Questionnaire SAQ-7 Physical limitation scale SAQ-7 angina stability scale SAQ-7 angina frequency scale SAQ-7 angina quality of life EQ-5D-5L Beck depression inventory

The SAQ-7 "angina frequency" domain has been shown to correlate to improvements in microvascular function in the WISE study. SAQ-7-7 has been also used in a number of studies, including the ISCHEMIA study.

Other patient questionnaires are also standardized tests for the assessment of quality of life, depression and symptom severity in coronary artery disease studies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and <85 years.
* Chronic coronary syndrome (including patients with anginal equivalents)
* Angina CCS class II-IV
* Evidence of reversible ischemia on non-invasive testing
* Availability of the following measurements:

  1. Index of microvascular resistances (IMR),
  2. Resting full-cycle ratio (RFR),
  3. Fractional flow reserve (FFR),
  4. Coronary flow reserve (CFR)
* Willingness to participate and ability to understand read and signed the informed consent document before the procedure

Exclusion Criteria:

At least one of the following:

* Pregnancy and or lactation.
* Medical or psychological conditions that would jeopardize an adequate and orderly participation.
* Left ventricular ejection fraction lower than 30%
* Previous coronary artery bypass surgery (CABG) to all major branches in the LAD and left circumflex (LCX) territory, such that IMR cannot be measured
* Decompensated congestive heart failure (CHF)
* Chronic or acute renal failure with creatinine >2mg/dl
* Severe valvular heart disease
* Patients with comorbidities limiting life expectancy to less than one year

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with angina without apparent obstructive coronary artery disease (no coronary stenosis >75% at angiography) undergoing clinically-indicated assessment of coronary microvascular function.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2029-10-10 (Estimated)

PRIMARY OUTCOMES:
Prognostic impact of resting resistances | 12 months
  The impact of resting resistances (expressed as Mean Transit Time, i.e. time for a saline bolus to reach the wire thermistor times distal pressure) on the incidence of patient-oriented outcomes (composite of cardiovascular death, myocardial infarction, rehospitalization for angina or heart failure and unplanned coronary angiography) at 12 months

SECONDARY OUTCOMES:
Correlation between SAQ measures and IMR | 6 months, 1 year and yearly to 5 years.
  Correlation of IMR with Seattle Angina Questionnaire, including each of its components (SAQ-7 Physical limitation scale, SAQ-7 angina stability scale, SAQ-7 angina frequency scale, SAQ-7 angina quality of life) at 6 months, 1 year and yearly to 5 years
Correlation between depression and IMR | 6 months, 1 year and yearly to 5 years.
  Correlation of IMR with Beck depression inventory scores
Correlation between physical ability and IMR | 6 months, 1 year and yearly to 5 years.
  Correlation of IMR with parameters of 5-EQ-EL
Distribution of mean transit time (Tmn) | At inclusion
  Distribution of Tmn (seconds).
Distribution of index of microvascular resistances (IMR) | At inclusion
  Distribution of IMR, units.
Distribution of aortic and distal pressure | At inclusion
  Distribution of Pa (aortic pressure) and Pd (distal arterial pressure) in mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsmedizin Mainz, Mainz, RLP, Germany

IPD SHARING:
Plan to Share IPD: No